CLINICAL TRIAL: NCT04063501
Title: Longitudinal Evaluation of Microbial and Host Signatures During Immunotherapy for Lung Cancer
Status: Recruiting | Type: Observational
Sponsor: NYU Langone Health (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 18-01845
Record Dates: First submitted 2019-08-19; First posted 2019-08-21 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-12

CONDITIONS: Lung Cancer
MeSH Terms: conditions — Lung Neoplasms | interventions — Bronchoscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Bacterial DNA will be extracted using an ion exchange column (Qiagen). Microbial DNA samples will potentially be further analyzed for relationships with underlying pathologies as well as to characterize in detail the genetic pool and genetic interactions..
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Advanced stage unresectable Non-Small Cell Lung Cancer: Adult patients with a diagnosis of advanced stage unresectable Non-Small Cell Lung Cancer and indication for PD-1 blockade treatment (either as monotherapy or combined with chemotherapy)
  Interventions: Other: Bronchoscopy; Other: Research Procedures

INTERVENTIONS:
Other: Bronchoscopy — The patient will then return within a week for a research bronchoscopy to sample the upper and lower airways
Other: Research Procedures — electrocardiogram, blood work (CBC, chemistry, coagulation profile and liver function tests, pregnancy test if applicable), X-ray and pulmonary function (spirometry) testing, and provide the patient with a stool collection kit.

SUMMARY:
This study will prospectively collect airway, stool, and blood samples on 80 subjects with lung cancer undergoing immunotherapy. Investigators will evaluate airway/stool microbial signatures associated with local (lower airway) and systemic (blood) immune tone.They will then study whether microbiota and/or host signatures predict subjects' response by longitudinal assessment of the progression free survival. They will also repeat sampling after 8 weeks of immunotherapy to expand our mechanistic understanding of the response to treatment.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with a diagnosis of advanced stage unresectable Non-Small Cell Lung Cancer and indication for PD-1 blockade treatment (either as monotherapy or combined with chemotherapy)

Exclusion Criteria:

* Antibiotic, steroid, or chemotherapy received within the prior month since these are possible confounders that may impact the microbiome and the host immunity.
* Brain metastasis (as evaluated by MRI obtained as part of standard of care staging evaluation)
* FEV1<50% predicted
* Cardiovascular disease (defined as abnormal EKG, known or suspected coronary artery disease or congestive heart failure)
* Renal disease
* Coagulopathy
* Liver disease

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with a diagnosis of advanced stage unresectable Non-Small Cell Lung Cancer and indication for PD-1 blockade treatment (either as monotherapy or combined with chemotherapy)
Sampling Method: Non-Probability Sample
Enrollment: 48 (Estimated)
Dates: Start 2021-02-09 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) | 3 Years
  over ≥ 1-year follow-up
Microbiota signatures in lower and upper airways | 3 Years
Microbiota signatures in stool | 3 Years

CONTACTS AND LOCATIONS:
Overall Officials: Leopoldo N Segal, MD, MSc, Principal Investigator — New York Langone Health
Locations (1):
- NYU Langone Health, New York, New York, United States